CLINICAL TRIAL: NCT03431311
Title: Protocol for Treatment Under Hospital Exemption: T Cell Receptor Based Therapy of Metastatic Colorectal Cancer With mRNA-engineered T Cells Targeting Transforming Growth Factor Beta Receptor Type II (TGFβII)
Brief Title: T Cell Receptor Based Therapy of Metastatic Colorectal Cancer
Acronym: TCR-CRC-001
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Svein Dueland, Principal Investigator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCR-CRC-001
Record Dates: First submitted 2018-01-30; First posted 2018-02-13 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Colorectal Cancer
Keywords: MSI
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adoptive Cell Therapy (ACT) (Experimental): The ACT will be administered as two intravenous (i.v.) injections of GMP TCR T cells per week for 6 weeks.
  Escalating dose per week, from 1 x108 cells (week 1) to 2x109 cells (week 4 onwards) using a central venous catheter. The doses listed indicate the maximum number of T cells per injection at any given time point.
  Interventions: Biological: Adoptive Cell Therapy (ACT)

INTERVENTIONS:
Biological: Adoptive Cell Therapy (ACT) — T cell receptor based therapy of metastatic colorectal cancer with mRNA-engineered T cells targeting mutant transforming growth factor beta receptor type II (TGFβII)

SUMMARY:
T Cell Receptor Based Therapy of Metastatic Colorectal Cancer With mRNA-engineered T Cells Targeting Transforming Growth Factor Beta Receptor Type II (TGFβII)

DETAILED DESCRIPTION:
Patients with advanced metastatic colorectal cancer who have no other effective treatment options will be offered the treatment. These patients have a poor prognosis, and there is a strong need for improved therapy.

The patients will be given adoptive cell therapy (ACT) with Radium-1 TCR+ T cells transiently redirected against the TGFβRII frameshift antigen which is expressed in MSI+ colon cancer. The first report on TCR therapy in colon cancer was targeting carcinoembryonic antigen (CEA) where some evidence of clinical response was seen, but the T-cell function may have been inhibited due to the necessity to resolve the severe colitis which occurred due to the presence of CEA in normal cells in the colon. This demonstrates the feasibility of T-cell therapy in metastatic colon cancer, but also the limitations of targeting CEA as an antigen.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic colon cancer which is MSI+ with the presence of the -1A deletion in TGFβRII gene, and positive for HLA-A02 genotype
* Measurable disease
* Female or male patients. Fertile females must have a negative pregnancy test before inclusion in the trial. Both fertile men and women must be ready and able to use highly effective methods of contraception, defined as use of oral, implanted, injectable, and mechanical or barrier products for the prevention of pregnancy during participation of the trial
* Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 1
* Age 18 years and older
* Life expectancy of at least 3 months
* Signed informed consent (by the subject or subject's legal representative) obtained before any trial-related procedures.
* Adequate organ function, measured by pre-defined laboratory values

Exclusion criteria

* Other metastatic malignancies
* Any other anti-tumour treatment within 4 weeks prior to first administration of cells.
* Steroid treatment, except substitution dose
* Significant cardiac or other medical illness that would limit activity or survival, such as severe congestive heart failure, unstable angina or serious cardiac arrhythmia
* Active infection requiring antibiotic therapy
* Pregnancy or lactation
* Known hypersensitivity to any of the components of the investigational product
* Patients who test positive for hepatitis B, C, HIV or syphilis
* Any reason why, in the opinion of the investigator, the patient should not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Incidence, nature, and severity of adverse events graded according to NCI CTCAE v4.0 | 2 years
  Incidence, nature, and severity of adverse events graded according to NCI CTCAE v4.0

SECONDARY OUTCOMES:
Progression free survival (PFS) | 2 years
  PFS defined as time from treatment to objective progression (as assessed by RECIST v1.1)
Radiological response rate (ORR) | 2 years
  ORR defined as the proportion of patients with an objective tumor response
Overall survival (OS) | 2 years
  OS defined as time from treatment to date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Svein Dueland, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway